CLINICAL TRIAL: NCT03416881
Title: Older HIV-infected Adults and Drug Interactions: Nationwide Cross-sectional Study Based on French National Health Insurance Databases
Brief Title: Older HIV-infected Adults and Drug Interactions: French Cross-sectional Study
Acronym: POPVIH65
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 1934895
Record Dates: First submitted 2017-11-09; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2017-11

CONDITIONS: HIV Infections
Keywords: HIV infection; antiretroviral; aging population; drug interactions; cross-sectional study; SNIIRAM
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Drug interactions between antiretroviral drugs and concomitants drugs and between antiretroviral need to be studied HIV-population is ageing. The referential of interactions is the Liverpool base.

DETAILED DESCRIPTION:
Filters in the French social security system database, 2016 :

* Code of Pathology "Human Immunodeficiency Virus (HIV) infection" Age ≥ 65 years
* Treatment with an antiretroviral between January 1, 2016 and December 31, 2016

ELIGIBILITY:
Inclusion Criteria:

* Men and women over than 65 years with an HIV infection and insured at the French Primary Health Insurance fund

No exclusion Criteria

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: French older HIV-infected adults (over than 65 years)
Sampling Method: Non-Probability Sample
Enrollment: 13225 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
frequency of major drug-drug interactions | between Jan, 1st 2016 and Dec, 31st 2016
  MDDI between 2 drugs (ARV/ARV or ARV/non-ARV) delivered during the same period yielding to a "Do Not Coadminister" statement, according to the University of Liverpool website (www.hiv-druginteractions.org/checker).

SECONDARY OUTCOMES:
costs associated with major drug-drug interactions | during 2016
  The costs were defined as all reimbursed healthcare acts recorded in the SNIIRAM